CLINICAL TRIAL: NCT00516295
Title: A Randomized Phase II Study of Bevacizumab (NSC 704865) Combined With Vincristine, Topotecan and Cyclophosphamide in Patients With First Recurrent Ewing Sarcoma
Brief Title: Vincristine Sulfate, Topotecan Hydrochloride, and Cyclophosphamide With or Without Bevacizumab in Treating Young Patients With Refractory or First Recurrent Extracranial Ewing Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00369; NCI-2009-00369 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AEWS0521 (Other: Children's Oncology Group); AEWS0521 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2007-08-14; First posted 2007-08-15 (Estimated); Results first posted 2014-09-02 (Estimated); Last update posted 2014-09-02 (Estimated); Status verified 2014-07

CONDITIONS: Ewing Sarcoma of Bone; Extraosseous Ewing Sarcoma; Peripheral Primitive Neuroectodermal Tumor; Recurrent Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor
MeSH Terms: conditions — Neuroectodermal Tumors, Primitive, Peripheral | interventions — Topotecan; trioctyl phosphine oxide; Vincristine; Cyclophosphamide; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (Feasibility assessment of VTCB) (Experimental): Patients receive bevacizumab IV over 30-90 minutes on day 1, vincristine sulfate IV on days 1, 8, and 15, and topotecan hydrochloride IV over 30 minutes and cyclophosphamide IV over 60 minutes on days 1-5. Treatment repeats every 21 days (except during weeks 14, 15 [course 5], 17, 18 [course 6], 26, 27 [course 9], 29, and 30 [course 10] when no chemotherapy is given) for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: topotecan hydrochloride; Drug: vincristine sulfate; Drug: cyclophosphamide; Biological: bevacizumab
- Arm II (VTCB) (Experimental): Patients receive bevacizumab, vincristine sulfate, topotecan hydrochloride, and cyclophosphamide as in Arm I.
  Interventions: Drug: topotecan hydrochloride; Drug: vincristine sulfate; Drug: cyclophosphamide; Biological: bevacizumab
- Arm III (CTC) (Active Comparator): Patients receive vincristine, topotecan hydrochloride, and cyclophosphamide as in arm I.
  Interventions: Drug: topotecan hydrochloride; Drug: vincristine sulfate; Drug: cyclophosphamide

INTERVENTIONS:
Drug: topotecan hydrochloride — Given IV
  Other Names: hycamptamine; Hycamtin; SKF S-104864-A; TOPO
Drug: vincristine sulfate — Given IV
  Other Names: leurocristine sulfate; VCR; Vincasar PFS
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
  Arms: Arm I (Feasibility assessment of VTCB); Arm II (VTCB)

SUMMARY:
This phase II trial study has a 6-patient feasibility portion studying the tolerability of chemotherapy with vincristine sulfate together with topotecan hydrochloride, cyclophosphamide, and bevacizumab in treating young patients with refractory or first recurrent extracranial Ewing's sarcoma. If the therapy is considered tolerable, this feasibility run-in will be followed by a randomized phase II portion studying giving vincristine sulfate together with topotecan hydrochloride, and cyclophosphamide to see how well it works compared with giving vincristine sulfate together with topotecan hydrochloride, cyclophosphamide, and bevacizumab in treating young patients with refractory or first recurrent extracranial Ewing's sarcoma. Drugs used in chemotherapy, such as vincristine sulfate, topotecan hydrochloride, and cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop tumor growth by blocking blood flow to the tumor. Giving combination chemotherapy together with bevacizumab may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of administering bevacizumab in combination with vincristine (vincristine sulfate), topotecan hydrochloride, and cyclophosphamide (VTC) to younger patients with refractory or first recurrent Ewing sarcoma.

II. To compare the progression-free survival of patients treated with VTC with bevacizumab vs VTC without bevacizumab.

SECONDARY OBJECTIVES:

I. To estimate the response rate to 2 cycles of VTC compared to 2 cycles of VTC/bevacizumab.

II. To evaluate biological markers as related to prognosis and specifically related to angiogenesis by encouraging concurrent enrollment on the Ewing sarcoma banking studies (COG-AEWS02B1 and/or COG-AEWS07B1) and ancillary correlative endothelial cell, surrogate marker, and angiogenic gene studies.

OUTLINE: This is a single therapy feasibility study followed by a randomized controlled portion. Patients are stratified according to time to disease recurrence (< 2 years vs >= 2 years).

ARM I (Feasibility assessment of VTCB): Patients receive bevacizumab intravenously (IV) over 30-90 minutes on day 1, vincristine sulfate IV on days 1, 8, and 15, and topotecan hydrochloride IV over 30 minutes and cyclophosphamide IV over 60 minutes on days 1-5. Treatment repeats every 21 days (except during weeks 14, 15 [course 5], 17, 18 [course 6], 26, 27 [course 9], 29, and 30 [course 10] when no chemotherapy is given) for up to 12 courses in the absence of disease progression or unacceptable toxicity.

ARM II (VTCB): Patients receive bevacizumab, vincristine sulfate, topotecan hydrochloride, and cyclophosphamide as in Arm I.

ARM III (VTC): Patients receive vincristine sulfate, topotecan hydrochloride, and cyclophosphamide as in arm I.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* ALT =< 5 times ULN for age
* Urine protein: creatinine ratio =< 0.5 OR 24-hour urine protein < 1,000 mg
* At least 6 weeks since other prior substantial bone marrow radiation
* At least 28 days since prior major surgical procedures (e.g., resection of tumor, laparotomy, thoracotomy, or open biopsy)
* At least 2 weeks since prior myelosuppressive chemotherapy (4 weeks for nitrosoureas)
* At least 2 weeks since prior local palliative radiotherapy (e.g., small port)
* Diagnosis of extracranial Ewing sarcoma or primitive neuroectodermal tumor of bone or soft tissue meeting 1 of the following criteria: I) a first recurrence of localized disease; II) a first recurrence of initially metastatic disease; III) disease refractory to initial conventional therapy
* Patients must have RECIST-measurable disease documented by clinical, radiographic, or histological criteria
* Patients who do not have measurable disease (e.g., bone scan-determined metastatic disease only) remain eligible for the study and will be evaluable for disease-free progression
* Karnofsky performance status (PS) 50-100% (> 16 years of age) OR Lansky PS 50-100% (=< 16 years of age )
* Life expectancy >= 8 weeks
* Absolute neutrophil count >= 1,000/μL
* NOTE: Patients with tumor metastatic to bone marrow are permitted to receive transfusions to maintain hemoglobin and platelet counts. These patients will not be evaluable for hematologic toxicity. Patients who are refractory to platelet infusions (i.e., unable to maintain platelet counts > 75,000/μL) and have marrow involvement and platelet counts < 75,000/μL are not eligible
* Fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy
* At least 1 week since prior therapy with a biologic agent or growth factor
* Patients must have histological verification of the malignancy at original diagnosis
* Histological confirmation of relapse is highly recommended but not mandatory
* Prior initial therapy with topotecan hydrochloride is allowed as long as > 2 years have elapsed since the initial diagnosis of Ewing sarcoma
* Prior therapy with cyclophosphamide or vincristine is allowed
* Minor surgical procedures (e.g., biopsies) for limited purposes of tissue retrieval allowed
* Minor procedures include indwelling IV catheter placement and needle biopsy for diagnostic purposes
* For minor surgeries, patients should not receive the first planned dose of bevacizumab until the wound is healed and 7 days have elapsed
* At least 6 months since prior craniospinal radiotherapy or radiotherapy to >= 50% of the pelvis
* At least 3 months since prior autologous stem cell transplantation (SCT)
* Platelet count >= 75,000/μL (transfusion independent)
* Hemoglobin >= 8.0 g/dL (may receive RBC transfusions)
* Direct bilirubin =< 1.5 times upper limit of normal (ULN) for age
* Creatinine clearance or radioisotope GFR >= 70 mL/min OR serum creatinine normal for age
* Hypertension must be well controlled on stable doses of medication for >= 2 weeks prior to enrollment
* Negative pregnancy test
* Female patients who are lactating must agree to stop breast-feeding
* II) The patient has no active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)
* Shortening fraction > 28% OR ejection fraction > 50%
* Recovered from any prior surgical procedure
* Sexually active patients of childbearing potential must agree to use effective contraception
* Patients on full-dose anticoagulants (e.g., warfarin) with PT INR > 1.5 are eligible if both of these criteria are met:
* I) The patient has an in-range INR (usually between 2 and 3) on a stable dose of oral anticoagulant or on a stable dose of low molecular weight heparin

Exclusion Criteria:

* Radiological or clinical evidence for parenchymal brain metastases or neuro axis involvement
* Documented, chronic nonhealing wound, ulcer, or significant traumatic injury (those with bone fractures, including pathological fractures, or requiring surgical intervention) within the past 28 days
* Other bone complications
* Deep venous thrombosis (including pulmonary embolism) within the past 3 months
* Recent (i.e., within 6 months) arterial thromboembolic events, including transient ischemic attack or cerebrovascular accident
* History of myocardial infarction, severe or unstable angina, or peripheral vascular disease Prior bevacizumab
* Radiotherapy or surgery for local control of recurrent disease concurrently with bevacizumab (bevacizumab must be held if radiotherapy or surgery is required)
* Radiotherapy to localized painful lesions is allowed, provided >= 1 measurable lesion is not irradiated
* Radiotherapy for local metastatic tumor control allowed after the first 2 courses of therapy
* Other cancer chemotherapy or immunomodulating agents
* Steroid use is allowed
* Prior allogeneic SCT

Ages: 1 Year to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2008-02; Primary Completion 2009-08 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Leavey, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Feasibility Assessment of VTCB) | Arm II (VTCB) | Arm III (CTC)
Started | 7 | 0 | 0
Completed | 4 | 0 | 0
Not Completed | 3 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — Ineligible | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm III (VTC): Patients receive vincristine sulfate, topotecan hydrochloride, and cyclophosphamide as in arm I.
- Total: Total of all reporting groups
Arm/Group | Arm I (Feasibility Assessment of VTCB) | Arm II (VTCB) | Arm III (VTC) | Total
Number analyzed (Participants) | 7 | 0 | 0 | 7
Age, Continuous [Median (Full Range); unit: years] | 15 [12 to 20] |  |  | 15 [12 to 20]
Gender [Number; unit: participants]
  Female | 2 |  |  | 2
  Male | 5 |  |  | 5
Race (NIH/OMB) [Number; unit: participants]
  American Indian or Alaska Native | 0 |  |  | 0
  Asian | 0 |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
  Black or African American | 0 |  |  | 0
  White | 6 |  |  | 6
  More than one race | 0 |  |  | 0
  Unknown or Not Reported | 1 |  |  | 1
Ethnicity (NIH/OMB) [Number; unit: participants]
  Hispanic or Latino | 2 |  |  | 2
  Not Hispanic or Latino | 5 |  |  | 5
  Unknown or Not Reported | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 |  |  | 7

OUTCOME MEASURES:

1. Primary Outcome: The Occurrence of Limiting Toxicity in an Eligible and Evaluable Patient.
Description: Limiting toxicity defined as Any Grade IV hematological toxicities lasting longer than 7 days, myelosuppression causing delays > 14 days in delivery of therapy, > Grade 3 thromboembolic events, > Grade 3 bleeding events, > Grade 2 hypertension, > Grade 2 proteinuria.
Time Frame: First 2 courses (42 days) of therapy
Population: Patients found not to meet the eligibility requirements are by group policy not followed for adverse events or outcome.
Measure: Number; unit: number of toxicities
Arm/Group | Arm I (Feasibility Assessment of VTCB) | Arm II (VTCB) | Arm III (VTC)
Number analyzed (Participants) | 6 | 0 | 0
number of toxicities | 0 |  |

2. Primary Outcome: Time to Disease Progression in Patients Receiving VTC With or Without Bevacizumab
Description: Time from enrollment to disease progression, death, second malignant neoplasm, or last patient follow-up whichever occurs first. Patients who experience disease progression, death or second malignant neoplasm will be considered to have experienced an event; otherwise the patient will be considered censored at last follow-up.
Time Frame: Maximum of 5 years after enrollment
Population: Patients found not to meet the eligibility requirements are by group policy not followed for adverse events or outcome.
Measure: Median (95% Confidence Interval); unit: days of event free survival
Arm/Group | Arm I (Feasibility Assessment of VTCB) | Arm II (VTCB) | Arm III (VTC)
Number analyzed (Participants) | 6 | 0 | 0
days of event free survival | 442 [42 to NA] — There is no numerical limit available because the limit is infinity. |  |

ADVERSE EVENTS:
Description: Patients found not to meet the eligibility requirements are by group policy not followed for adverse events or outcome.
Arm/Group | Arm I (Feasibility Assessment of VTCB) | Arm II (VTCB) | Arm III (VTC)
Serious Adverse Events (participants affected / at risk) | 5/6 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 6/6 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Feasibility Assessment of VTCB) (N=6) | Arm II (VTCB) (N=0) | Arm III (VTC) (N=0)
Burn (Injury, poisoning and procedural complications) | 1 | 0 (0) | 0
Esophageal stenosis (Gastrointestinal disorders) | 1 | 0 (0) | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 0 (0) | 0
Infections and infestations - Other, specify (Infections and infestations) | 4 | 0 (0) | 0
Platelet count decreased (Investigations) | 1 | 0 (0) | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 (0) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Feasibility Assessment of VTCB) (N=6) | Arm II (VTCB) (N=0) | Arm III (VTC) (N=0)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Allergic reaction (Immune system disorders) | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 6 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Catheter related infection (Infections and infestations) | 1 | 0 | 0
Creatinine increased (Investigations) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Esophageal infection (Infections and infestations) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 2 | 0 | 0
Lymphocyte count decreased (Investigations) | 2 | 0 | 0
Middle ear inflammation (Ear and labyrinth disorders) | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 4 | 0 | 0
Oral hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 2 | 0 | 0
Platelet count decreased (Investigations) | 4 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0 | 0
White blood cell decreased (Investigations) | 3 | 0 | 0

LIMITATIONS AND CAVEATS:
In preparing to re-open for randomized enrollment in November, 2008 the study committee was asked to amend the study and the decision was made to close AEWS0521 for administrative purpose.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less